CLINICAL TRIAL: NCT05777226
Title: Multi-center Study of Natural History of SORD-related Charcot-Marie-Tooth Disease and Epalrestat Treatment
Brief Title: Research of SORD-CMT Natural History and Epalrestat Treatment
Acronym: SORD-CMT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Ruxu Zhang, Director, Chief physician of Neurology, The Third Xiangya Hospital of Central South University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: quick22474
Record Dates: First submitted 2023-02-13; First posted 2023-03-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Charcot-Marie-Tooth Disease (CMT)
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — epalrestat; Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epalrestat treatment group (Experimental): Epalrestat;Tablet; 50mg; three times a day; 36 months
  Interventions: Drug: Epalrestat
- control group (No Intervention): No Intervention

INTERVENTIONS:
Drug: Epalrestat — Patients in the treatment group are intervened with Epalrestat tablets.
  Other Names: Epalrestat Tablets（YANGTZE River Pharmaceutical Group Nanjing Pharmaceutical. Co., Ltd.）
  Arms: Epalrestat treatment group

SUMMARY:
Charcot-Marie-Tooth disease (CMT) is a group of the most common hereditary peripheral neuropathy with high clinical and genetic heterogeneity. Biallelic pathogenic variants in SORD gene leading to loss of function of SORD protein cause axonal degeneration. Current research suggests that SORD-CMT2 may be the most common subtype of AR-CMT2. The primary purpose of this study is to explore the natural history of SORD-CMT2 patients by detecting the ONLS scale score and serum sorbitol level changes at 6th, 12th, 24th, and 36th months and to evaluate the effectiveness and safety of epalrestat. Patients with strong treatment willingness and voluntary purchase of drugs are included in the epalrestat treatment group, and patients without drug treatment willingness are included in the control group. Patients in the drug treatment group take epalrestat (50 mg) orally three times daily. This study is expected to be carried out simultaneously in 5 hospitals in mainland China. About 30 SORD-CMT2 patients will be enrolled in this study, and the study period will be 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed SORD-CMT2 patients.
* Male or non-pregnant, non-lactating female patients, aged > 14 and ≤ 50 years old.
* Rule out secondary peripheral neuropathy (e.g., diabetic peripheral neuropathy)
* Voluntarily participate in clinical trials, sign informed consent, and be able to understand and abide by research procedures.

P.S. Patients who have a strong willingness to treat and voluntarily purchase epalrestat for treatment (50mg, three times a day) are included in the treatment group.

Exclusion Criteria:

* Presence of any other cause of peripheral neuropathy.
* Subjects with other neurological disorders affecting the evaluation of study treatment.
* History of clinically significant unstable medical disease that may cause harm to subjects participating in this study within the past 1 year.
* Patients with major trauma or extremity surgery before enrollment or planned for extremity surgery before completion of follow-up.
* Patients with previous bilateral ankle stabilization surgery.
* Patients who were treated with other related drugs in the 3 months before enrollment.
* Have any history of drug abuse; have a history of alcohol dependence in the past 3 months.
* Subjects who are positive for syphilis antibody and HIV antibody.
* Subjects whose chest X-ray and B-ultrasound show tumors.
* Patients with poor compliance and unable to complete the study follow-up.
* Patients who do not agree to participate in the study.
* Other factors are not suitable for inclusion.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Serum sorbitol levels | 36 months
  Changes of serum sorbitol levels at 6, 12, 24 and 36 months
Overall Neuropathy Limitations Scale (ONLS) scores | 36 months
  Changes in ONLS scale scores at 6, 12, 24, and 36 months, The total score for the arm is 5 points and 7 for the leg; the total score ranges from 0 points (no disability) to 12 points (disability)

SECONDARY OUTCOMES:
The 10-meter walk test (10MWRT) | 36 months
  Changes in the 10-meter walk test (10MWRT) at 6, 12, 24, and 36 months

IPD SHARING:
Plan to Share IPD: No